CLINICAL TRIAL: NCT05224440
Title: Partnered Implementation Evaluation of a National Sponsorship Program for Transitioning Service Members ( PEC 20-170)
Brief Title: National Sponsorship Program for Transitioning Service Members
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Central Texas Veterans Health Care System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: PEX 21-001; 1I50HX003258-01A1 (NIH)
Record Dates: First submitted 2022-01-10; First posted 2022-02-04 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Reintegration Difficulties; Health; Suicidal Ideation and Behaviors; Connectedness
Keywords: Reintegration difficulties; Transitioning Servicemember/Veteran; Veteran Sponsorship Initiative; Connectedness; Suicide prevention; VA Utilization; Community intervention; Stepped Wedge
MeSH Terms: conditions — Suicidal Ideation; Behavior; Suicide Prevention

STUDY DESIGN:
Intervention Model Description: To execute the Hybrid Type 2, we will use a stepped wedge design, which relies on sequential roll-out to participating cities over time. The cities in Texas with the largest population density of veterans were selected. Our design also enables us to make efficient use of all data available for within-site and between-site comparisons. The comparison examines cities as they cross-over from Transition as Usual (TAU) to intervention. The between-site comparison evaluates the intervention period for a city vs. all other intervention and TAU periods for all cities. We randomized at the city level and will use TSMVs as the unit of observation for primary quantitative outcome measures. Six cities are participating in the evaluation, with two cities allocated to each of the three start dates or steps. Because cities differ regarding organizational characteristics, we used the restricted selection method of randomization to balance cities based on the number of projected TSMV moving to target.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Veteran Sponsorship Initiative (Experimental): TSMV receives a VA certified and volunteer sponsor (1-on-1) approximately 6 months prior to military discharge. Sponsorship continues for approximately 6 months after military discharge.
  Interventions: Behavioral: Veteran Sponsorship Initiative
- Transition as Usual (No Intervention): TSMVs transition to civilian life as usual.

INTERVENTIONS:
Behavioral: Veteran Sponsorship Initiative — Consistent with preventive, universal and public health approaches to suicide, the VA's TSMV Sponsorship Initiative establishes public-private partnerships with federal and community organizations to provide TSMVs with one-on-one, certified and volunteer sponsors in their post-military hometowns. Sponsors are assigned approximately six months prior to discharge and help TSMVs to accomplish reintegration tasks pre-and post-discharge. After certification, sponsors are assigned to and managed by a community integration coordinator (CIC), which is a local organization. CICs recruit sponsors, manage sponsors and match sponsors with TSMVs moving to the local region. After being matched with a TSMV, sponsors then integrate their skills during regular contact with matched TSMVs and monthly video or in-person sessions and help TSMVs identify SMART goals and develop reintegration action plans and ensure TSMVs attend VA healthcare appointments.
  Arms: Veteran Sponsorship Initiative

SUMMARY:
Background:

The United States is undergoing a suicide epidemic for its youngest Veterans (18-to-34-years-old) as their suicide rate has almost doubled since 2001. Veterans are at the highest risk during their first-year post-discharge, thus creating a "deadly gap" for them. In response, the nation has developed strategies that emphasize a preventive, universal and public health approach and embrace the value of community interventions. The three-step theory of suicide suggests that community interventions that reduce pain from reintegration difficulties and promote connectedness for Veterans as they transition to civilian life have the greatest likelihood of success. Recent research shows that the effectiveness of community interventions can be enhanced when augmented by volunteer and certified sponsors (1-on-1) who actively engage with Veterans, as part of the Veterans Affairs' Transitioning Servicemember/Veteran (TSMV) Sponsorship Initiative.

Method/Design:

The purpose of this trial is to determine how to implement the Veteran Sponsorship Initiative in six cities in Texas in collaboration with the US Department of Defense, VA, Texas government, and local stakeholders. Texas is an optimal location for this large-scale implementation as it has the second largest population of Veterans aged 18-to-34-years-old and is home to the largest US military installation, Fort Hood. The first aim is to further determine the effectiveness of the Sponsorship Initiative, as evidenced by measures of proximal variables (reintegration difficulties, health/psychological distress, VA healthcare utilization and connectedness) and distal variables (suicidal ideation and behaviors). The second aim is to determine how best to implement the Veteran Sponsorship Initiative in Texas with the intent of future expansion in more states. TSMVs (n=630) will be recruited from military installations six months prior to discharge and prior to moving to target cities. The evaluators are utilizing implementation strategies, such as building community partnerships and external facilitation. Evaluation will be conducted through interviews with TSMVs and periodic reflections with key stakeholders to identify barriers, facilitators, and adaptations. Outcome evaluations will be conducted with TSMVs completing surveys and data collection from working with stakeholders.

Discussion:

This evaluation will have important implications for the national implementation of community interventions that address the epidemic of TSMV suicide. Aligned with the Evidence Act, it is the first large-scale implementation of an evidence-based practice that conducts a thorough assessment of TSMVs during the "deadly gap".

DETAILED DESCRIPTION:
The United States is undergoing a suicide epidemic for its youngest Veterans (18-to-34-years-old) as their suicide rate has almost doubled from 23.62 suicide deaths per 100,000 in 2001 to 44.44 per 100,000 in 2019. Their current rate is 1.65 times higher than older Veterans and 2.73 times higher than non-Veterans of the same age. The approximately 200k Servicemembers that exit the active-duty military every year are at the highest risk for suicide during their first-year post-discharge as the rate almost triples during this period and remains elevated for up to six years. Therefore, the period between discharge and successfully reintegrating into civilian life is a "deadly gap". Traditional and clinical approaches offered by the VA to address the epidemic have been limited as only 24% of active-duty SMs that exit the military per year enroll in VA healthcare within the first-year post-discharge. And when servicemembers (SMs) and Veterans do seek healthcare services or are assessed for suicide risk, about 70% of them who later attempt suicide deny suicidal ideation in the months leading up to their suicide attempt.

In response, the White House developed a recent strategy that emphasizes a preventive and public health approach and embraces the value of public-private partnerships with community organizations to reduce SM and veteran suicide. Aligned with the White House's strategy, the VA has similarly implemented a public health approach that emphasizes proactive community interventions. Their intent is to implement more universal and preventive interventions that are upstream to address social determinants of health and risk factors for suicide (e.g., lack of connectedness, financial concerns/unemployment, relationship distress). Recent national legislation supports the focus on community interventions as the Commander John Scott Hannon Act will provide $174 million to organizations that provide community interventions which address suicide risk factors and engage with Veterans not participating in VA clinical care.

Klonsky and May's three-step theory of suicide (3ST) provides a theoretical basis for such preventive, universal and public health approaches to suicide that emphasize community interventions for transitioning servicemembers and Veterans (TSMVs). The primary tenants of the 3ST are that (a) suicidal ideation results from a combination of pain, primarily psychological pain, and hopelessness, (b) connectedness is a key protective factor against increasing suicidal ideation, and (c) progression from suicide ideation to attempt occurs when factors create sufficiently high capacity to end one's life.

For TSMVs, psychological pain can be attributed to reintegration difficulties. Sokol and colleagues describe how reintegration difficulties for TSMVs can be a pervasive source of pain that create the first step towards suicidal ideation. Many TSMVs report high levels of reintegration difficulties, particularly related to education/employment, housing, food security, health, relationship challenges and legal involvement. Civilian employment is often cited as a significant concern as 43 percent of SMs are not fully prepared nor career-ready as they exit the military. And as they enter the civilian workforce many TSMVs struggle to translate their military skillsets into a civilian setting with TSMVs changing jobs twice within the first three years of transition.

The reintegration difficulties that TSMVs experience can persist for over 6 years and indeed contribute to increased suicide risk. In fact, Kline and colleagues found that 45% of SMs endorse difficulties post-discharge and that those with the highest number of difficulties are at 5.42 times greater risk of suicidal ideation. Overall, it appears that reducing reintegration difficulties is likely to be a critical component of community interventions that prevent suicide.

Based on the 3ST, the second critical component of community interventions is likely to be promoting connectedness for TSMVs. Klonsky and colleague highlight that connectedness most often means connection to other people but can also refer to an attachment to a job, project, role, interest, or any sense of perceived purpose or meaning that keeps one invested in living. The military goes to great lengths to promote connectedness throughout a SM's career by providing them specially selected and trained leaders to assist them (e.g., recruiters, drill sergeants, and unit leaders) with these leaders being held accountable for the welfare of each assigned SM. The individualized support continues as SMs train with their units and deploy to combat with research showing that positive leadership has a beneficial effect on the mental health of combatants.

Even prior to conducting a permanent change of station (PCS) and moving from one military installation to another, the military provides all SMs with a PCS sponsor. For instance, the U.S. Marine Corps has a thorough and required PCS sponsorship program that intends to reduce stress and challenges associated with relocating. PCS Sponsors are of equal rank and matched based on gender, marital status, and career field. They orient their matched SMs to their new installation and help them accomplish their transition tasks. The support received from such leaders is considered critical for SMs to accomplish their designed mission within the military.

Though, as TSMVs exit the military and attempt to reintegrate to their civilian life they experience a dearth of support from the military in their post-military hometowns. The same recruiter that was there to enlist them into the military is not there to assist in their reintegration. Additionally, when TSMVs return home, there are far fewer individuals, employers, family members and colleagues with whom they can relate. Therefore, it is not surprising that TSMVs report that they feel closer to their military comrades than to their civilian counterparts after exiting the military.

VA's Veteran Sponsorship Initiative There is a growing body of research showing mentorship/sponsorship interventions may potentially benefit TSMVs. Eby and colleagues conducted a meta-analysis of 112 studies, primarily with non-TSMVs, and found that mentoring is associated with favorable relational, career and mental health outcomes. Specific to the VA's TSMV Sponsorship Initiative, Geraci and colleagues conducted a 3-arm randomized controlled trial (n=200) and used hierarchical linear modeling to assess the impact of community interventions with TSMVs being assessed at baseline, 3-months, 6-months and 12-months. The results showed the limitations of some community interventions to reduce reintegration difficulties and improve connectedness for TSMVs. Importantly, it also showed that the effectiveness of community interventions can be enhanced when augmented by the Sponsorship Initiative, especially with the Expiration Term of Service Sponsorship Program. It also highlighted that TSMVs who rated their sponsors as high for task-oriented (e.g., "emphasizes the meeting of deadlines") and relational-oriented (e.g., "is friendly and approachable") leadership behaviors had significantly reduced reintegration difficulties compared to TSMVs who rated their sponsors as low.

Since establishment of the Foundations for Evidence-based Policymaking Act (Evidence Act., US PL 115-435) of 2018, VA must use evidence and evaluation to inform policies and budget allocations. Therefore, the current evaluation has important implications for the national implementation of community interventions that address the epidemic of TSMV suicide. This evaluation is the first large-scale implementation of an evidence-based practice that conducts a thorough assessment of TSMVs during the "deadly gap".

This project is jointly funded by VA leadership within Texas and the VA Quality Enhancement Research Initiative (QUERI) through a peer-reviewed Partnered Evaluation Initiative (PEI) grant. The PEI grants are one of the VA's principal methods to meet the requirements of the Evidence Act and focus on improving veteran health by rapidly implementing evidence-based practices and planning for national scale-up and spread. Texas has the second largest population of Veterans aged 18 to 34 years old, which makes it an ideal state for a large-scale implementation of the Sponsorship Initiative.

Study Aims The purpose of this Hybrid Type 2 effectiveness-implementation evaluation is to expand upon previous work that established the evidence base for the Veteran Sponsorship Initiative to determine how to implement the initiative in major metropolitan regions of Texas in collaboration with the US Department of Defense, VA, Texas government, and local stakeholders. The first aim is to further determine the effectiveness of the Sponsorship Initiative, as evidenced by measures of proximal variables (reintegration difficulties, health/ psychological distress, VA health service utilization and connectedness) and distal variables (suicidal ideation and behaviors). The second aim is to determine the feasibility and potential utility of implementing the Sponsorship Initiative in six cities in Texas (Austin, San Antonio, Houston, Dallas/Fort Worth, El Paso, and Corpus Christi) with the intent of developing processes and a toolkit to facilitate future expansion in more states. The third aim is to determine the effectiveness of the Sponsorship Initiative, as evidenced by change scores in the same outcome for the first aim, for TSMVs identified as high risk for suicide.

TSMV Participants and Recruitment TSMVs will be recruited into the Veteran Sponsorship Initiative using targeted outreach at participating military installations. They will be informed of the Sponsorship Initiative during mandatory Transition Assistance Program classes that TSMVs must attend prior to military discharge and encouraged to register for the Sponsorship Initiative through the ETS-SP website. To be eligible for enrollment, TSMVs must be 18-years of age or older, be approximately 6 months from military discharge and be planning to transition to one of the target cities included in the evaluation during an active enrollment window for the respective city. The first 315 TSMVs that enroll will be assigned to the TAU group; the next 315 TSMVs per step will be assigned to the Sponsorship Initiative.

To determine necessary sample size needed for this evaluation, statistical power analysis was completed using the powerlmm package (Magnusson, 2018) within the R computing environment. To test the primary hypothesis, that the Sponsorship Initiative reduces reintegration difficulties (as assessed by the M2C-Q) with power of 80%, alpha of .05, and moderate effect size (partial eta squared of .06) between the TAU and Sponsorship Initiative groups, the total number of TSMVs to be enrolled across the six cities is 630. This sample size allows for adjustments required under randomization, design effects, and expected attrition of approximately 30% between enrollment and the final post-military discharge assessment.

Potential sponsors will be recruited in target cities using social media outreach with the local VA, Veteran Service Organizations, and college and university alumni networks. In accordance with previous research, the investigators anticipate a sponsor attrition rate of approximately 20%. Therefore, to mitigate the risk of developing a shortage of sponsors, the sponsorship initiative aims to recruit a sufficient number of sponsors to ensure a 1-on-1 capacity for TSMVs.

Analyses Hierarchical models will be used to analyze quantitative data. TSMVs will be nested within each city when analyzing data collected during the specified timepoints. Hierarchical random effects models examine within- and between-group change across time and by group (TAU vs. Sponsorship Initiative). The investigators will use mixed effects modeling as it accounts for the underlying heterogeneity between and within participants (i.e., intercepts and slopes are allowed to vary across participants). This approach will also allow us to identify differences in rates of change (slopes) in the dependent variables between groups and to control for confounding variables that may influence TSMV outcomes (e.g., gender). Hierarchical models incorporate participants with missing data by estimating the best fitting model from the data available for each participant. Therefore, for the intent-to-treat (ITT) analyses all data points for TSMVs who conduct the pre-implementation assessment will be entered into the model.

During the qualitative interviews, near-verbatim notes from TSMV interviews and periodic reflections with partners will be uploaded and maintained in Atlas.ti qualitative software, allowing for qualitative and mixed-method analyses. Qualitative thematic analysis will then be used to identify the most frequently mentioned areas.

Discussion As suicide rates for the youngest Veterans, especially for those during their first-year post-discharge, continue to increase national efforts have recently emphasized preventive, universal and public health approaches that embrace the value of public-private partnerships with community organizations to reduce SM and veteran suicide. As identified in the 3ST, community interventions that reduce pain associated with reintegration difficulties and improve connectedness have the potential to reduce TSMV suicidal risk. By partnering with organizations already serving TSMVs, it is possible that national suicide prevention efforts will be more effective. Recent research shows that this effectiveness can be enhanced when augmented by sponsors who actively engage with TSMVs, such as in the Sponsorship Initiative.

This evaluation will have important implications for the national implementation of community interventions that address the epidemic of TSMV suicide. Aligned with the Evidence Act, it is the first large-scale implementation of an evidence-based practice that conducts a thorough assessment of TSMVs during the "deadly gap". The study protocol described in this manuscript-a Hybrid Type 2 implementation-effectiveness evaluation-was developed in close partnership with relevant operations partners and will use state-of-the-art evaluation methods to answer key questions regarding how best to implement and sustain initiatives such as the Veteran Sponsorship Initiative. Specifically, mixed quantitative and qualitative data collection will allow the investigators to develop clear guidance for operations partners regarding context-sensitive implementation strategies to address multi-level barriers to initiative implementation and sustainment. Results will also contribute to knowledge of how reintegration difficulties can be understood across multiple locations, which is vital to ensuring effective processes and generalizable results across sites.

ELIGIBILITY:
Inclusion Criteria:

* TSMVs must be 18-years of age or older,
* be approximately 6 months from military discharge and
* be planning to transition to one of the target cities included in the evaluation during an active enrollment window for the respective city.

Exclusion Criteria:

N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 630 (Estimated)
Dates: Start 2022-02-04 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Military to Civilian Questionnaire (M2C-Q; Sayer et al., 2011) | Change in baseline scores across 4 timepoints [ Time Frame: Baseline, 4 months after, 8 months after, 12 months after]
  Reintegration difficulties will be assessed using the Military to Civilian Questionnaire (Primary Outcome; M2C-Q; Sayer et al., 2011), a 16-item measure that assesses reintegration difficulties in (a) interpersonal relationships with family, friends, and peers; (b) productivity at work, in school, or at home, (c) community participation; (d) self-care; (e) leisure, and (f) perceived meaning in life. Items are rated on a 5-point Likert scale ranging from 0 (No difficulty) to 4 (Extreme difficulty). Minimum: 0 (best); Maximum: 4 (worst)

SECONDARY OUTCOMES:
Employment/education status | Change in baseline scores across 4 timepoints [ Time Frame: Baseline, 4 months after, 8 months after, 12 months after]
  Employment/education status will be assessed by asking TSMVs to self-report if they are currently enrolled as a student in any educational institute, and their current work status. If they are not a student nor employed, then the TSMV is asked "What have you been doing in the past 4 weeks to find work?".
Brief Resilience Scale (BRS; Smith et al., 2008) | Change in baseline scores across 2 timepoints [ Time Frame: Baseline and 12 months after]
  Resilience will be assessed using the Brief Resilience Scale (BRS; Smith et al., 2008), a 6-item scale with strong evidence of validity, test-retest reliability, and internal consistency across samples (Windle et al., 2011). One of the questions is: "I tend to bounce back quickly after hard times". Items are rated on a 5-point Likert scale ranging from 1 (Strongly Disagree) to 5 (Strongly Agree). Minimum:1 (worst); Maximum: 5 (best)
VA Homelessness Screening Clinical Reminder (HSCR; Montgomery, 2014) | Change in baseline scores across 2 timepoints [ Time Frame: Baseline and 12 months after]
  Homelessness will be assessed using the VA Homelessness Screening Clinical Reminder (HSCR; Montgomery, 2014), a four-item measure that assesses current homelessness or imminent risk of homelessness among Veterans. The HSCR is considered a standard of care within VA settings to identify and respond to instances of Veteran homelessness. One of the questions is: "In the past two months, have you been living in stable housing that you own, rent, or stay in as part of a household?" A "No" response indicates the TSMV is positive for homelessness.
U.S. Adult Food Security Survey Module (2012) | Change in baseline scores across 2 timepoints [ Time Frame: Baseline and 12 months after]
  Food insecurity will be assessed using the U.S. Adult Food Security Survey Module (2012), a three-stage screening measure for assessing food insecurity. An example question is: "Within the past 12 months, the food that I bought just didn't last, and I didn't have money to get more". A response of "often" or "sometimes" is an indication that the TSMV is experiencing food insecurity.
Criminal behaviors | Change in baseline scores across 2 timepoints [ Time Frame: Baseline and 12 months after]
  Criminal behaviors are assessed using a series of self-report items, including "Within the last 12 months have you been issued a ticket of any kind for a traffic violation (e.g., speeding, failure to signal)?"; "Within the last 12 months have you been arrested or charged for any type of criminal offense (e.g., DUI, disorderly conduct, drug offense, domestic violence, assault, robbery)?"; and "Within the last 12 months, has a restraining order, no contact agreement, or order of protection been initiated or taken against you?"
Well-Being Signs | Change in baseline scores across 2 timepoints [ Time Frame: Baseline and 12 months after]
  Well-Being Signs is a three-item screening measure, based on the work of Vogt et al. (2021) used to assess how TSMVs are doing in their daily lives. It asks TSMVs to rate what percentage of time (from 0 to 100%) that they have been "Fully satisfied with how things are going in these aspects of life?", "Regularly involved in all aspects of life that are important to you?", and "Functioning your best in aspects of life that you do participate in?". Minimum: 0% (worst); Maximum: 100% (best)
VA healthcare enrollment and utilization | Change in baseline scores across 4 timepoints [ Time Frame: Baseline, 4 months after, 8 months after, 12 months after]
  VA healthcare enrollment and utilization will be assessed through the VA Corporate Data Warehouse (CDW), which enables us to access data for TSVMs who have enrolled and utilized VA healthcare services. Vanneman et al. (2015) conducted one of the first studies to identify predictors of VA enrollment and utilization for TSMVs. Importantly, they identified that there was a three-fold increase in VA enrollment and utilization during the first-year post-discharge for TSMVs who engaged in VA healthcare services prior to discharge. Therefore, this evaluation will begin the enrollment process early for TSMVs while they are still within the military.
Generalized Anxiety Disorder Questionnaire (GAD-7; Spitzer et al., 2006) | Change in baseline scores across 4 timepoints [ Time Frame: Baseline, 4 months after, 8 months after, 12 months after]
  Symptoms of anxiety will be assessed using the Generalized Anxiety Disorder Questionnaire (GAD-7; Spitzer et al., 2006). The GAD-7 is a 7-item self-report scale routinely used in primary care settings as a psychometrically sound screener for clinically significant anxiety (Jordan et al., 2017). Minimum: 0 (best); Maximum: 21 (worst)
Patient Health Questionnaire-9 (PHQ-9; Kroenke et al., 2010) | Change in baseline scores across 4 timepoints [ Time Frame: Baseline, 4 months after, 8 months after, 12 months after]
  Depression will be assessed using the Patient Health Questionnaire-9 (PHQ-9; Kroenke et al., 2010), a 9-item self-report measure that has shown strong construct validity, test-retest reliability, and internal reliability across samples (Kroenke et al., 2010; Corson et al., 2004; Currier et al., 2015). Minimum: 0 (best); Maximum: 27 (worst)
Primary Care PTSD 5 (PC-PTSD-5; Prins, et al., 2016) | Change in baseline scores across 4 timepoints [ Time Frame: Baseline, 4 months after, 8 months after, 12 months after]
  Symptoms of posttraumatic stress will be assessed using the Primary Care PTSD 5 (PC-PTSD-5; Prins, et al., 2016), a brief, self-report scale that shows excellent utility as a psychometrically sound screener for clinically significant posttraumatic stress disorder in military Veterans (Prins et al., 2016). Minimum: 0 (best); Maximum: 5 (worst)
Alcohol Use Disorders Identification Test-Consumption (AUDIT-C; Bush, et al., 1998) | Change in baseline scores across 4 timepoints [ Time Frame: Baseline, 4 months after, 8 months after, 12 months after]
  At-risk drinking behaviors will be assessed using the Alcohol Use Disorders Identification Test-Consumption (AUDIT-C; Bush, et al., 1998), a three-item, psychometrically strong, screening measure for alcohol misuse. The AUDIT-C is routinely used within VA settings to screen outpatients for at-risk drinking behaviors. Minimum: 0 (best); Maximum: 12 (worst)
Somatic symptom burden will be assessed by the Somatic Symptom Scale 8 (SSS-8; Gierk, et al., 2014) | Change in baseline scores across 4 timepoints [ Time Frame: Baseline, 4 months after, 8 months after, 12 months after]
  Somatic symptom burden related to stomach problems, back pain, headaches, chest pain, dizziness, energy, and sleep will be assessed by the Somatic Symptom Scale 8 (SSS-8; Gierk, et al., 2014). Previous studies with Veterans demonstrated good item characteristics and excellent reliability, a sound factor structure and significant associations with related constructs like depression, anxiety, pain, quality of life and impairment (Toussaint et al., 2017)
Medical Outcomes Study Social Support Survey (MOS-SSS; Sherbourne & Stewart, 1991) | Change in baseline scores across 4 timepoints [ Time Frame: Baseline, 4 months after, 8 months after, 12 months after]
  Connectedness will be assessed using the Medical Outcomes Study Social Support Survey (MOS-SSS; Sherbourne & Stewart, 1991), a 19-item self-report measure of perceived availability of social support or connectedness that has demonstrated strong psychometric properties in military (Erbes et al., 2017), Veteran (Currier et al., 2013; Tsai et al., 2020), and civilian samples (Sherbourne & Stewart, 1991). Minimum: 1 (worst); Maximum: 5 (best)
Columbia-Suicide Severity Rating Scale (C-SSRS) screener (Posner et al., 2011) | Change in baseline scores across 2 timepoints [ Time Frame: Baseline and 12 months after]
  Risk for suicidal ideation and behaviors will be assessed using procedures described by Katz et al. (2019). The VA Intake team will ask questions from the Columbia-Suicide Severity Rating Scale (C-SSRS) screener (Posner et al., 2011) supplemented by questions based on cues provided in the full C-SSRS about suicide attempts ("Have you attempted suicide or done harm to yourself or put yourself in a dangerous situation with the intent of ending your life"), and about injuries ("Did it result in you needing to get medical care with a doctor or hospital"). TSMVs will be placed in hierarchical categories based on their highest level of reported ideation or behavior. Minimum: 0 (best); Maximum: 7 (worst)
Reach | Change in baseline percentages across 4 timepoints for each military installation [Time Frame: Initiation of evaluation for each military installation, 4 months after, 8 months after, and 12 months after]
  Reach will be assessed by calculating the percent of eligible TSMVs that sign up for the Sponsorship Initiative compared to the total number of eligible TSMVs on respective military installations.
Adoption (Sponsors) | Change in baseline percentages across 4 timepoints for each city [Time Frame: Initiation of evaluation for each city, 4 months after, 8 months after, and 12 months after]
  Adoption will be assessed by the percent of sponsors who sign up for the Sponsorship Initiative and then become certified.
Maintenance (number of sponsors) | Change in numbers across 2 timepoints for each city [Time Frame: 12 months after initiation of evaluation for each city and 6 months after)
  Maintenance (number of sponsors) will be evaluated after the implementation phase and operationalized as the number of sponsors engaged with the sponsorship initiative.
Income status | Change in baseline scores across 4 timepoints [ Time Frame: Baseline, 4 months after, 8 months after, 12 months after]
  Income status will be assessed by asking TSMVs to self-report total combined income, including spouse and family, and the amount of money they have set aside in case of an unexpected financial events.
Maintenance (number of CICs) | Change in numbers across 2 timepoints for each city [Time Frame: 12 months after initiation of evaluation for each city and 6 months after)
  Maintenance (number of CICs) will be evaluated after the implementation phase and operationalized as the number of CICs engaged with the sponsorship initiative.
Maintenance (number of TSMVs) | Change in numbers across 2 timepoints for each city [Time Frame: 12 months after initiation of evaluation for each city and 6 months after)
  Maintenance (number of TSMVs) will be evaluated after the implementation phase and operationalized as the number of TSMVs engaged with the sponsorship initiative.
Maintenance (VA funding) | Change in funding across 2 timepoints for each city [Time Frame: 12 months after initiation of evaluation for each city and 6 months after)
  Maintenance (VA funding) will be evaluated after the implementation phase and operationalized as the amount of funding dedicated to the sustainment and expansion of the sponsorship initiative.
Implementation (Quality of delivery) | One timepoint [Time Frame: 12 months after Baseline]
  Implementation (Quality of delivery). TSMV evaluation of sponsor through the Leader-Behavior-Description-Questionnaire-LBDQ (Halpin, 1957).
Level of personality functioning will be assessed by the Level of Personality Functioning Scale-Brief Form 2.0 (Weekers et al. 2018) | Change in baseline scores across 4 timepoints [ Time Frame: Baseline, 4 months after, 8 months after, 12 months after]
  Level of personality functioning will be assessed by the Level of Personality Functioning Scale-Brief Form 2.0 (Weekers et al. 2018), which serves as a quick assessment of personality dysfunction severity as defined by Criterion A of the DSM-5 Alternative Model for Personality Disorders. It captures features of self-pathology, including poor self-worth and affective instability, which have close relationships with self-reported suicidality (Bach et al., 2020).
Implementation (Participant responsiveness: Completion of "My Action Plan") | Change in percentages across 4 timepoints for each city [Time Frame: Initiation of evaluation for each city, 4 months after, 8 months after, and 12 months after]
  Implementation (Participant responsiveness: Completion of "My Action Plan"). Will be measured by the percent of the initial "My Action Plan" completed by TSMVs with their sponsors.
Adoption (Community Integration Coordinators) | Change in baseline number across 4 timepoints for each city [Time Frame: Initiation of evaluation for each city, 4 months after, 8 months after, and 12 months after]
  Adoption (Community Integration Coordinators) will be calculated by the number of CICs who become actively involved and sign a VA Memorandum of Agreement.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph C Geraci, PhD, Principal Investigator — James J. Peters Veterans Affairs Medical Center
Locations (2):
- United States (2):
  - James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York
  - Central Texas Veterans Health Care System Waco VA Medical Center, Waco, TX, Waco, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Geraci JC, Finley EP, Edwards ER, Frankfurt S, Kurz AS, Kamdar N, Vanneman ME, Lopoo LM, Patnaik H, Yoon J, Armstrong N, Greene AL, Cantor G, Wrobleski J, Young E, Goldsmith M, Seim RW, Goodman M. Partnered implementation of the veteran sponsorship initiative: protocol for a randomized hybrid type 2 effectiveness-implementation trial. Implement Sci. 2022 Jul 8;17(1):43. doi: 10.1186/s13012-022-01212-9. PMID 35804354